CLINICAL TRIAL: NCT03098576
Title: Personalized Cancer Care at Cedars-Sinai Medical Center Samuel Oschin Comprehensive Cancer Institute
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Monica Mita, Associate Professor of Medicine, Cedars-Sinai Medical Center
Other Study IDs: IIT2015-20-Mita-CSMCMatch
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cancer
Keywords: advanced; metastatic solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh or archived tissue Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Matched: Matched targeted drug treatment
  Interventions: Other: Matched targeted drug treatment
- Control: Unmatched standard of care
  Interventions: Other: Unmatched standard of care

INTERVENTIONS:
Other: Matched targeted drug treatment — Matching a specific genetic abnormality (i.e. mutation) with the appropriate targeted drug.
  Groups: Matched
Other: Unmatched standard of care — All patients with either no identified mutation or no available matching treatment but undergoing a systemic treatment will be enrolled in the "control group."
  Groups: Control

SUMMARY:
The purpose of this study is to examine the usefulness of matching patients to targeted therapy by analyzing a tumor sample taken at diagnosis and testing it against 50 cancer-associated genes. Targeted therapy is a highly personalized, newer approach to cancer treatment that aims to more precisely identify and attack cancer cells, in an effort to do less damage to normal cells.

DETAILED DESCRIPTION:
Targeted therapy in this study can be either off label-use of a U.S. Food and Drug Administration (FDA) approved drug or a clinical trial that includes investigational drugs. Matched targeted therapy outcomes will be compared to the outcomes of patients who were not matched to a treatment.

In order to find a matched treatment, a patient's sample will undergo a test known as a "gene chip algorithm." This is will be done by having a sample of a patient's tumor analyzed at a Cedars-Sinai Medical Center (CSMC) laboratory that specializes in molecular profiling. Molecular profiling is a process used to study a tumor's genetic characteristics. DNA will be taken from the tumor sample and will be screened for "actionable genes." These genes are called actionable because mutations (structural changes) in these genes have FDA-approved matched therapies or are eligible for current clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Advanced and metastatic solid tumors who have failed standard treatments known to improve survival
* Female and male adults age 18 and older.
* ECOG PS 0-2
* Acceptable hematological, renal, or liver function
* Patients planning to undergo a systemic treatment
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Significant comorbidities that could interfere with the study (compliance and visits)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced and metastatic solid tumors who have failed standard systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 years
  To evaluate the proportion of patients with response to targeted study agent(s) in patients with advanced cancers.

SECONDARY OUTCOMES:
Progression free survival | 6 months
  To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced cancers.
Overall survival | 3 years
  Evaluate time until death.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Mita, MD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No